CLINICAL TRIAL: NCT07078266
Title: Multicenter Comparative Study on the Diagnostic Efficacy of "Ultra-high Sensitivity" Cardiomagnetic Detection and Myocardial Nucleoradiology Scanning for Early Diagnosis of Myocardial Ischemia.
Brief Title: Comparative Study of Magnetocardiography and Emission Computed Tomography.
Status: Not yet recruiting | Type: Observational
Sponsor: Yang Jing (Other)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Yang Jing, Associate Researcher, Chongqing Emergency Medical Center
Organization: Chongqing Emergency Medical Center (Other)
Other Study IDs: 2025-28
Record Dates: First submitted 2025-06-24; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Myocardial Ischemia
Keywords: Coronary atherosclerotic Heart Disease; Coronary Microvascular Disease; Myocardial Ischemia; Magnetocardiograph; Emission Computed Tomography
MeSH Terms: conditions — Myocardial Ischemia; Microvascular Angina

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Magnetocardiography examination — Magnetocardiography (MCG) is a non-invasive, risk-free, and contactless technology that characterizes the local magnetic field signals generated by the electrical activity of the heart.
  the magnetic signals used in magnetocardiograms can pass through the body with almost no interference. Therefore, magnetocardiography theoretically offers more clinically useful information, with the advantages of being non-invasive, safe, and fast, enabling earlier and more accurate diagnoses of potential heart diseases.

SUMMARY:
Coronary atherosclerotic heart disease (CHD) and Coronary Microvascular Disease (CMVD), as the primary etiologies of myocardial ischemia, have garnered increasing clinical attention due to their high prevalence and severe prognostic implications.

Currently, the primary method for detecting myocardial ischemia is Emission Computed Tomography (ECT). However, it suffers from limitations such as low spatial resolution and radiation exposure risks.magnetocardiography(MCG) is a non-invasive, contactless medical imaging device that maps localized magnetic signals generated by cardiac electrical activity.The magnetocardiography (MCG) system constructs cardiac magnetic field images by recording biomagnetic signals via a multi-channel sensor array positioned above the thoracic region.MCGcan capture the spatial magnetic field changes of ischemic myocardial cells, and carry out early warning, early diagnosis and positioning detection of myocardial ischemia.

This study is a prospective, multicenter, controlled trial. The study will enroll adult patients presenting with myocardial ischemia symptoms suspected of having coronary heart disease (CHD) or coronary microvascular disease (CMVD), who are scheduled to undergo ECT examination.and a domestically manufactured "ultra-high sensitivity" cardiomagnetic detection device will be used to collect cardiac magnetic images. The ECT examination will be completed within one week. A consistency analysis will be conducted between the cardiac magnetic results and the ECT results to evaluate the early diagnostic efficacy of cardiac magnetic detection for myocardial ischemia. Subgroup analyses will also be performed based on resting and stress conditions.

Primary study endpoints:Diagnostic Performance of MCG in Detecting Myocardial Ischemia: Positive Predictive Value, Specificity, and Sensitivity.

Secondary study endpoint:Concordance and Discrepancies Between MCG and ECT in Diagnosing Myocardial Ischemia.

DETAILED DESCRIPTION:
1. Research Background Magnetocardiography (MCG) is a non-invasive, risk-free, and contactless technology that characterizes the local magnetic field signals generated by the electrical activity of the heart. The magnetic signals from the heart and the electrical signals from the heart are of the same origin. The ionic activity within myocardial cells forms volume currents, and the curve representing the potential difference caused by these currents on the body surface over time is known as the Electrocardiogram (ECG). The spatial magnetic field changes caused by volume currents are referred to as magnetocardiograms. Magnetocardiograms are constructed by recording the magnetic signals of the heart using a multi-channel sensor array placed above the chest, thereby mapping the heart's magnetic field. By analyzing these magnetic maps, abnormal electrical activities of the heart can be detected, including myocardial ischemia, arrhythmias, and myocardial diseases. Traditional ECG detection technology is affected by various conductivities of human tissues and skin, whereas the magnetic signals used in magnetocardiograms can pass through the body with almost no interference. Therefore, magnetocardiography theoretically offers more clinically useful information, with the advantages of being non-invasive, safe, and fast, enabling earlier and more accurate diagnoses of potential heart diseases.Earlier magnetocardiography (MCG) systems were not adopted clinically because of their prohibitive costs and technical challenges.Recently,our country has successfully developed a heart magnetic measurement device based on spin-exchange relaxation-free magnetic measurement technology. This device has successfully completed 64-channel time-sharing heart magnetometry and 32-channel synchronous heart magnetometry.The core component of the heart magnetic detection device is the SERF atomic magnetometer, which uses a novel alkali metal atom operating in the SERF state to achieve extremely weak magnetic measurements. It has advantages such as non-cryogenic operation (traditional magnetometers require cooling with liquid helium), miniaturization, and high spatial resolution.The basic principle is: using high temperature to achieve a higher density of alkali metal vapor in the gas cell, suppressing spin-exchange relaxation, and using polarized detection light that is perpendicular to the pump light entering the gas cell to measure the Larmor precession frequency of spin-polarized atoms in a weak magnetic field, thus accurately reflecting the magnitude of the external magnetic field. The SERF magnetometer has achieved high sensitivity to low-frequency magnetic fields in weak magnetic fields.Therefore, MCG device can ultra-sensitively, non-invasively, and dynamically display human cardiac magnetic functional information, reflecting corresponding electrophysiological activities of the heart. It provides a novel tool for the clinical diagnosis and evaluation of cardiovascular diseases, holding broad application prospects in medicine.
2. Research Objectives This study aims to compare the domestically developed "ultra-sensitive" MCG device with ECT, the gold standard for myocardial ischemia detection, to determine whether the domestic "ultra-sensitive" MCG device can accurately identify myocardial ischemia, thereby exploring its clinical application value.
3. study design This study is a prospective, multi-center comparative study. 3.1 research contents 3.1.1 Recruit participants and collect data Patients who come to our hospital for treatment with myocardial ischemia symptoms such as chest tightness and chest pain and plan to undergo ECT will be informed by the receiving doctor of the clinical study. Patients who are willing to participate in the study will be further communicated with the patient by the investigator to evaluate and confirm whether they meet the inclusion conditions, and inform that the study will collect clinical diagnosis and treatment information such as basic conditions, medical history, laboratory examinations, as well as study-related precautions, and sign informed consent form.

3.1.2 Preparation before magnetic examination Before undergoing magnetic electrocardiogram, the patient's basic information was asked and checked, the past history, alcohol and tobacco status, and the current medical history (the onset time, inducement, symptom characteristics, duration, etc. of chest pain) were recorded, and the subject's blood pressure, height, and weight were measured.

3.1.3 Magnetocardiography and ECT examination MCG images were collected using a domestic "ultra-high-sensitive" MCG detection device, and ECG examinations were performed 10 minutes before and after. ECT examination was completed within 1 week.

3.1.4 Data Entry The subject's diagnostic results, myocardial damage markers, heart failure indicators, electrocardiogram, echocardiography, coronary CTA/angiography, ECT and other laboratory test results were recorded and entered into EDC.

3.2 Data Analysis The consistency of Magnetocardiographic results and ECT results was analyzed to evaluate the effectiveness of magnetocardiographic testing in early diagnosis of myocardial ischemia.

3.3 Sample size Estimation In this project sample size calculation was performed to ensure the statistical reliability of the study. By considering factors such as the expected effect size and significance level, an appropriate sample size was determined. This ensures sufficient support for testing the study hypothesis, guarantees scientifically credible results, enhances study reproducibility, and boosts data analysis robustness, thereby making the study conclusions more convincing and reliable.

For testing the non - inferiority of cardiomagnetic evaluation of myocardial ischemia compared to ECT, the sample size estimation used the method for comparing paired two - sample rates in a non - inferiority design and was calculated as follows:

n=(Zα+Zβ)2×(p1(1-p1)+p2(1-p2))/(p1-p2-Δ)2 In the formula： Zα is the critical value of the standard normal distribution; Zβ is the critical value of the standard normal distribution corresponding to the power; P1 and P2 represent the positive rates of the control group and the intervention group, respectively; Δ：non-inferiority margin; α：significance level; β：power of the test. The preliminary experimental results indicated a 77% positive rate for cardiomagnetic detection and 71% for ECT， with α=0.05 (one - sided), β=0.2 (power 80%), and Δ=0.05. We calculated the minimum sample size to be 196 cases, with a total sample size of 196 cases. Considering a dropout rate of 10%, the final determined sample size was 218 cases.

3.4 Statistical Methods Unless otherwise stated, the following general principles will be used for statistical analysis of the study data.

For categorical variables, statistical descriptions will be provided as the number and percentage of participants in each category. For continuous variables, the mean, standard deviation, median, Q1，Q3 and extremes will be listed. Diagnostic efficiency will be evaluated using sensitivity, specificity, AUC, recall, and F1 score for discrimination. Calibration will be assessed via calibration curves and the Hosmer-Lemeshow (H-L) test. Subgroup analyses will be conducted for rest ECT and stress ECT groups to compare diagnostic efficiency and consistency. The Pearson correlation coefficient will assess the linear relationship between cardiomagnetic scores and ECT ischemic areas, with the correlation coefficient (r) and significance level (p value) reported. The Kappa coefficient will evaluate the consistency of cardiomagnetic detection with rest and stress ECT in diagnosing myocardial ischemia, with the consistency level reported.

All statistical tests will use a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Presence of myocardial ischemia-related symptoms (e.g., angina pectoris) with suspected CHD or CMVD, scheduled for ECT examination
* Signed informed consent form

Exclusion Criteria:

* Hemodynamic instability (systolic blood pressure <90 mmHg or requiring vasoactive drugs);
* Cardiac arrhythmias, including ventricular tachycardia, ventricular fibrillation, severe sinus bradycardia and sinus pauses, and second - degree or higher - degree atrioventricular block and other severe arrhythmias;
* Aortic dissection aneurysm, severe aortic valve stenosis or insufficiency;
* Elderly or frail patients with neuromuscular or osteoarticular diseases who cannot complete exercise stress ECT; Allergy to drugs used in pharmacologic stress ECT;
* Patients with severe renal insufficiency with an estimated glomerular 6.filtration rate (eGFR) < 30 ml/min or those undergoing dialysis;
* Patients with malignant tumors and a life - expectancy of less than1 year;
* Pregnant or lactating women;
* Patients unable to undergo MCG examination due to inability to enter the chamber, metallic implant interference, or other conditions deemed unsuitable by researchers.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will enroll adult patients presenting with myocardial ischemia symptoms suspected of having coronary heart disease (CHD) or coronary microvascular disease (CMVD), who are scheduled to undergo ECT examination.
Sampling Method: Probability Sample
Enrollment: 218 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation Indicators: Diagnostic concordance between " ultra-high sensitivity" magnetocardiography (MCG) and rest/stress ECT (including exercise and pharmacological stress protocols) for detecting myocardial ischemia. | 2025.7-2026.7

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT07078266/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT07078266/ICF_001.pdf